CLINICAL TRIAL: NCT02265575
Title: Hylenex-Assisted Resuscitation in Kenya (HARK) Trial for the Management of Dehydration
Acronym: HARK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brett D. Nelson, MD, MPH, DTM&H, Assistant Pediatrician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001390
Record Dates: First submitted 2014-10-07; First posted 2014-10-16 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — Hyaluronic Acid; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hyaluronic acid (Experimental): Rehydration using hyaluronidase-assisted subcutaneous infusion
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Hyaluronic Acid — rehydration using hyaluronidase-assisted subcutaneous infusion
  Other Names: hyaluronidase; Hylenex

SUMMARY:
One of the leading health issues among patients, particularly children, presenting for care in low- and middle-income countries is dehydration. When oral rehydration is not sufficient or is clinically inappropriate, rehydration often occurs intravenously. An alternative to intravenous rehydration is subcutaneous infusion and - with or without hyaluronidase enzyme (or Hylenex) - has been shown in several robust trials in high-income countries to be as effective and even safer than intravenous infusion. In this study in western Kenya, the investigators propose a first-ever randomized controlled trial to evaluate whether hyaluronidase-facilitated subcutaneous infusion can be as effective and safe as IV therapy among moderate-to-severely dehydrated patients in low- and middle-income countries.

DETAILED DESCRIPTION:
Subcutaneous (SC) infusion has been established in high-income countries as a safe and effective alternative to expedite and simplify IV access. , A study from 2003 demonstrated the efficacy of SC hydration in elderly patients, for example. Fluid absorption via the SC method was almost identical to that via the IV method. A recent retrospective study compared SC fluid infusion with IV fluid infusion in children and showed that the SC method makes possible a more timely delivery of parenteral fluid with fewer needlesticks.

Additionally, SC hydration has been shown to be even more effective with the addition of recombinant human hyaluronidase, an enzyme that breaks down hyaluronic acid that makes up the extracellular matrix. , (Note: Hyaluronidase, or Hylenex, is not an investigational drug; it is FDA-approved, regularly used in the U.S., and will be procured for this study through the pharmacy of the Massachusetts General Hospital (Boston, USA).) When hyaluronidase is injected subcutaneously, an area forms where fluids do not have a dense matrix to cross. Flow rates with hyaluronidase-assisted SC (hSC) infusion are nearly five times faster than SC fluid administration alone.8 U.S.-based studies comparing hSC rehydration with standard IV rehydration in children with mild-to-moderate dehydration have demonstrated several benefits of hSC, including time and success of line placement, ease of use, satisfaction, and cost-effectiveness.9, These studies concluded that hSC hydration is a reasonable alternative to IV hydration in resource-rich settings, especially for children with difficult IV access.

While hSC infusion has been shown to be safe, successful, and cost-effective in high-income countries like the United States, there have been no randomized control trials in low-resource settings. The benefits of hSC that have been demonstrated in high-income countries, namely the ease of use and cost-effectiveness, may be particularly advantageous in low- and middle-income countries. It may even be found to be safer in these settings than current standards of care in light of recent findings of higher mortality with IV bolus rehydration among febrile children with infection in Africa. We, therefore, propose a feasibility study to evaluate whether hSC infusion can be effective and safe among moderate-to-severely dehydrated patients in rural community hospitals in western Kenya.

Rationale

hSC infusion can improve clinical management of patients presenting with moderate-to-severe dehydration. It can serve as a definitive alternative rehydration method or as a bridge to IV access when IV access is unobtainable.

Hypotheses

Hyaluronidase-assisted subcutaneous fluid resuscitation is equally effective as standard IV therapy for initial volume resuscitation in moderate to severely dehydrated patients in rural Kenya.

Hyaluronidase-assisted subcutaneous fluid resuscitation can decrease costs, shorten time to IV placement (reduce needlesticks), less discomfort, and decrease complications compared to standard IV therapy in moderate to severely dehydrated patients in rural Kenya.

Research questions

This study seeks to help answer the following research questions: Can hSC be effectively introduced among mid-level providers in rural community hospitals in western Kenya? Can hSC serve as an effective and safe treatment or bridge to IV access among patients presenting with moderate-to-severe dehydration? What are the perceptions and attitudes of providers and patients upon the use of hSC? What is the cost effectiveness of hSC in this setting?

Objectives

To evaluate the efficacy of hyaluronidase-assisted subcutaneous resuscitation (hSC) in moderate to severely dehydrated patients in Kenya.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to a participating facility with moderate-to-severe dehydration will be considered for participation. Other inclusion criteria will include:
* Patients over the age of 1 month
* Patients presenting with moderate-to-severe dehydration who failed to improve or are not candidates for oral rehydration therapy and IV access is not successful twice
* Parents or legal guardian(s) available to provide written informed consent

Exclusion Criteria:

* There will be no limitation based on race, tribe, language, or sexual orientation in the study for any patients who meet treatment criteria. There are no exclusions based on language. Exclusion criteria will include:
* Any condition precluding SC infusion or infusion-site evaluation in all possible anatomic locations, including the upper back, anterior thighs, abdomen, and other potential areas for hSC therapy
* Any reason (before study enrollment) for a hospital admission or extended stay for other than dehydration-related illness
* Known hypersensitivity to hyaluronidase or any ingredient in the study formulation of recombinant human hyaluronidase
* Any patient not eligible for IV or SC fluids as determined by the local clinician
* Any medical condition likely to interfere with the patient's ability to fully complete all protocol-specified interventions, the ability to undergo all protocol-specified assessments, or likely to prolong the patient's need for medical attention beyond that required for addressing the dehydration-related illness

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to recovery | participants will be followed for the duration of hospital stay, an expected average of 3 days
  Time to normal fluid hydration status

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | participants will be followed for the duration of hospital stay, an expected average of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Brett D. Nelson, MD,MPH,DTM&H, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Sagam Community Hospital, Luanda, Kenya

REFERENCES:
- [Result] Zubairi H, Nelson BD, Tulshian P, Fredricks K, Altawil Z, Mireles S, Odongo F, Burke TF. Hyaluronidase-Assisted Resuscitation in Kenya for Severely Dehydrated Children. Pediatr Emerg Care. 2019 Oct;35(10):692-695. doi: 10.1097/PEC.0000000000001183. PMID 28678057